CLINICAL TRIAL: NCT02841839
Title: A Pilot Study to Evaluate Sampling Methods for Subgingival Plaque
Brief Title: A Study to Evaluate Sampling Methods for Subgingival Plaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016135
Record Dates: First submitted 2016-07-11; First posted 2016-07-22 (Estimated); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Subgingival Plaque
MeSH Terms: interventions — Tin Fluorides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2-step system (Experimental): Subjects are to brush with 2-step system for 4 weeks; stannous fluoride
  Interventions: Drug: Stannous Fluoride

INTERVENTIONS:
Drug: Stannous Fluoride

SUMMARY:
To identify a sampling method for collecting subgingival plaque

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study;
* Be 18 years of age or older;
* Agree not to participate in any other oral/dental product studies during the course of this study;
* Agree to delay any elective dentistry (including dental prophylaxis) until the study has been completed;
* Agree to use the acclimation toothpaste together with their regular brush and refrain from any other oral care products (including floss and mouth rinse) between the Screening and Baseline Visit;
* Agree to use the treatment products and refrain from any form of non-specified oral hygiene during the treatment periods (after the Baseline Visit), including but not limited to the use of products such as floss, mouth rinse, or whitening products;
* Agree to return for all scheduled visits and follow study procedures;
* Must have at least 16 natural teeth;
* Be in good general health, as determined by the Investigator/designee based on a review of the health history/update for participation in the study;
* Agree to refrain from all oral hygiene for at least 12 hours prior to each visit;
* Agree to refrain from eating, chewing gum, drinking and using tobacco for 4 hours prior to each visit;
* Have 10-20 bleeding sites; and
* Have minimum 6 sampling sites with bleeding and pocket depth ≥2mm but not deeper than 4mm.

Exclusion Criteria:

* Have had a dental prophylaxis within 2 weeks of plaque sampling visits;
* Have taken antibiotics or used anti-gingivitis / anti-bacterial oral care products such as chlorhexidine or Listerine within 2 weeks of plaque sampling visits;
* Have rampant caries, open or untreated caries, or advanced periodontitis requiring prompt treatment;
* Taking allergy medication or any other medication that can affect salivary flow such as an antihistamine;
* Need an antibiotic prophylaxis prior to dental visits;
* A history of hypersensitivity to oral care products containing hydrogen peroxide or stannous fluoride;
* A history of hypersensitivity to products containing sodium lauryl sulfate (SLS);
* Are pregnant (Self-reported) or lactating; or
* Have any condition or disease, as determined by the Investigator/Designee based on a review of the medical history, which could be expected to interfere with examination procedures or with the subject's safe completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Subgingival plaque | 4 weeks
  subgingival plaque quantity measured by periopaper or curette sampling